CLINICAL TRIAL: NCT05743543
Title: A Feasibility Study of a Sphenopalatine Ganglion (SPG) Block for Post Traumatic Stress Disorder (PTSD)
Brief Title: A Pilot Study of SPG Block for PTSD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Diana Martinez, Clinical professor in Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8104
Record Dates: First submitted 2023-01-31; First posted 2023-02-24 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active SPG block (Experimental): The block will be performed using a topical aerosolized nasal spray followed by the administration of a local anesthetic.
  Interventions: Other: Sphenopalatine ganglion block

INTERVENTIONS:
Other: Sphenopalatine ganglion block — The block is performed with a nasoscope and the administration of a local anesthetic.

SUMMARY:
Some patients with Post Traumatic Stress Disorder (PTSD) respond only partially to medication. This study is a pilot study investigating whether blocking the SPG helps reduce the symptoms of PTSD. This study does not involve treatment with medications. It is a proof of principal study.

DETAILED DESCRIPTION:
The sphenopalatine ganglion (SPG) is a collection of neurons involved in autonomic regulation (which refers to bodily processes that are automatic like heart rate and blood pressure). Blocking the SPG is used to treat disorders, such as migraines or cluster headaches (short, severe headaches that occur together). The procedure will be performed by a doctor who specializes in ear, nose throat surgery. The block consists of the injection of a numbing agent (similar to the type used by dentists) to the SPG. After the SPG block, we will follow patients for 8 weeks to see how they feel.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a principal diagnosis of PTSD on stable dose of psychiatric medication or in stable psychotherapy for at least 3 months, who experience residual symptoms.
* Participants who understand all study procedures and can undergo informed consent

Exclusion Criteria:

* Participants with a medical disorder, for whom study participation could be deleterious (neurologic, cardiac, renal or infectious disease)
* Pregnant or breast feeding participants
* Participants who are on an anticoagulant, such as warfarin, or otherwise have a medical condition that increases bleeding risk

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
feasibility: number of participants completing the 8-week study | 8 weeks
  feasibility: number of participants completing the 8-week study
tolerability: number of adverse events | 8 weeks
  tolerability: number of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- NYSPI, New York, New York, United States